CLINICAL TRIAL: NCT03024606
Title: Smoking Cessation Following Text Message Intervention in Pregnant Women
Brief Title: Smoking Cessation Intervention in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Katherine Mathews, MD, Principal Investigator, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23943
Record Dates: First submitted 2017-01-13; First posted 2017-01-19 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- texting group (Active Comparator): text messages focused on smoking cessation and pregnancy
  Interventions: Behavioral: text messages focused on smoking cessation and pregnancy
- control group (No Intervention): No text messages

INTERVENTIONS:
Behavioral: text messages focused on smoking cessation and pregnancy — The impact of a text-message service on smoking cessation in medically underserved, obstetric patients when added to the usual care of pharmacist-driven CBT smoking cessation program and smoking cessation pharmacotherapy with either the nicotine replacement patch or bupropion.
  Arms: texting group

SUMMARY:
The investigators propose an 18-month, randomized, open-label evaluation of the impact of texting to pregnant, underserved, cigarette smokers on smoking cessation rates. Patients will be eligible if they have a confirmed pregnancy, are English speaking, at least 18 years of age, are in the preparation stage of change and willing to set a quit date within 30 days and before 35 weeks gestation, and have a cellular phone that is capable of receiving text messages. Patients will be randomized to either the texting group or control group. A baseline carbon monoxide level will be obtained. The patient, regardless of group, will have the standard of care smoking cessation visit. If the pharmacist, physician, and patient deem that pharmacotherapy is appropriate, patient will receive nicotine replacement therapy patches or bupropion free of charge in 2-week intervals. Patients in the intervention group will receive text messages focused on smoking cessation and pregnancy. Patients will be seen on a bi-weekly schedule to obtain additional vouchers for patches or for bupropion, meet with the pharmacist, and complete a carbon monoxide exhalation test. These visits will be continued until the pharmacotherapy course is complete.

DETAILED DESCRIPTION:
Smoking during pregnancy has been shown to have detrimental effects on both the mother and the fetus. The perinatal period presents a critical opportunity to educate and support the mother as she attempts quit. Current studies suggest a median quit rate of only 4.9% in women receiving usual care (Cognitive Behavioral Therapy, CBT), but a number of studies have investigated new interventions in addition to usual care to help increase compliance with smoking cessation. Pharmacological aids such as nicotine replacement therapy (NRT) and bupropion are recommended as potential options by the American College of Obstetrics and Gynecology since they are considered safer than continued smoking during pregnancy. Studies thus far on smoking cessation with the help of electronic devices have demonstrated mixed results; however, the impact of texting in the pregnant population in combination with CBT and pharmacological therapy has yet to be assessed.

Smoking during pregnancy has been shown to have detrimental effects on both the mother and the fetus. Cigarettes contain over 3000 compounds many of which can cause risk to pregnancy. However, the nicotine and carbon monoxide components are of primary concern. Nicotine releases epinephrine, which results in a decrease in uterine blood flow and an increase in uterine resistance. There is also decreased production of fetal nitric oxide resulting in lower blood flow to the fetus and leading to decreased birth weight, length, and head circumference compared to non-smokers.

Studies have proven that exposure to tobacco can increase the risk for placental abruption, placental previa, preterm birth, antenatal death, sudden infant death syndromes, attention-deficit/hyperactivity disorder and asthma. Compared to children of non-smoking mothers, children of mothers who smoked during pregnancy had a higher BMI and increased odds for being overweight at 4-years of age; however, in the children whose mother quit smoking during pregnancy there was no increased risk of increased BMI or being overweight compared to the children of non-smoking mothers. According to the data from the 2009 Pregnancy Risk Assessment and Monitoring System (PRAMS) approximately 12.4% of pregnant women with live births reported smoking during the last three months of pregnancy (PRAMS). Of the 25% of women who smoked in the 3 months prior to pregnancy, 52% quit during pregnancy; of those, 44% relapsed within 6 months after delivery. The perinatal period presents a critical opportunity to educate and support the mother as she attempts quit.

Current studies evaluating rates of smoking cessation in pregnant women show less than ideal results. A primary analysis of 12 pooled trials found a median quit rate of 4.9% in women with usual care. This rate increased to 13.2% in patients that received tailored self-help intervention.12 To help increase compliance with cessation, studies have investigated new interventions as part of the usual care provided to pregnant patients that continue to smoke. One study looked at including a 15-minute video and provider prompting at baseline and one month. Although a higher percentage of patients in the intervention group had a higher 30-day abstinence rate at 2-months post baseline, the finding was not significant (26.1% vs 10.5%, p=0.12) although the study did not discuss if this was an appropriately powered sample size. Another study looking at the combination of smoking cessation education, physical activity counseling and supervised exercise found a 25% abstinence rate at 8-months gestation. The use of NRT has also been studied. One study found that CBT plus NRT verses CBT alone was effective at 7-weeks (24% vs 8%, p=0.02) and 38-weeks' gestation (18% vs 7%, p=0.04), unfortunately there was no benefit at 3-months post-partum (20% vs. 14%, p=0.55).

The use of pharmacological aids for smoking cessation is recommended as a potential option by the American College of Obstetrics and Gynecology. Currently, NRT products and bupropion are appropriate options during pregnancy and are the most utilized therapy for cessation during pregnancy. Although classified as pregnancy category-D medication, NRT patches are often used to assist the pregnant patient in smoking cessation when CBT is not successful. A review looking at 4-studies that examined pregnancy outcomes after NRT, found a significant decrease in the risk of preterm delivery and low-birth weight compared to active smokers. NRT is considered safer than continued smoking since it only provides nicotine whereas smoking provides nicotine plus over 3000 other chemicals. It has also improved cessation rates near the quit date compared to CBT in obstetric patients. Similarly, bupropion has improved cessation rates in non-obstetric patients and has not been associated with malformations or abnormal pregnancy outcomes.

The transtheoretical stages of change assessment is beneficial to help determine a patient's readiness to quit. Data has shown that the stages predict preparation for cessation and successful cessation. In the precontemplative stage, patients are not willing to consider smoking cessation. The contemplative stage is defined as patients considering smoking cessation but not ready to set a quit date. Preparation stage occurs when patient is ready to set a quit date within the next 30 days. In the action stage, patients have been smoke free for less than six months. Maintenance stage is cessation longer than 6 months. Relapse is when patients have starting smoking again after being in the action stage. In other obstetric smoking cessation literature, relapse has been defined as smoking more than 5 cigarettes or smoking more than 5 times since cessation.

Mobile technology is common place in today's society. According to the 2013 Nielsen report, 94% of all Americans 16 years of age or older use a cellular phone with more than half of those being smart phones. A total of 96% of phone owners have a data plan included. In 2012, the average monthly usage included 164.5 calls, 644.1 voice minutes, and 764.2 text messages. Ownership of cell phones and high tech devices extends to all socioeconomic classes, and the ease and affordability has made cell phone use common for all races and income brackets. When looking at text message specifically for race 79% of whites, 85% of Blacks and 87% of Hispanics report text messaging. When looking at household income 78% of those making < 30K, 80% of those making between 30k-50k, and 88% of those making greater than 50k are active texters. African Americans are more likely than the general population to own smart phones (71% vs. 62%) and are 44% more likely than the broader market to create a social media profile. Over a monthly basis, African Americans also spend 24% more time on their phone , 12% more time on email, and 10% more time on the internet. Hispanics text the greatest of all ethnic groups at 943 text messages per month. Based on this data, it is apparent that mobile phone messaging is a potential convenient and cost-effective way to interact with patients of all races and income levels.

Results of current studies looking at smoking cessation with the help of computer or other electronic device are mixed. Several trials have looked at the use of text-messaging based smoking cessation programs. One randomized controlled pilot trial of 151 daily smokers interested in quitting found a non-clinically significant difference in cessation rates at 3 months between the intervention and control groups (11% versus 4%), this study was not powered to detect a statistical difference. A small pilot study evaluating Text2Quit, an automated, personalized, and interactive program that sends texts and emails over the course of 3 months, reported liking the program at 2 and 4 weeks after enrollment (91% and 82%, respectively) and 75% of participants reported reading most or all of the messages sent. Unfortunately, the majority of participants admitted to smoking at the 4-week visit. The txt2stop study was a trial of 5800 smokers that were randomized to receive text messages that were comprised of motivational and behaviour-change support versus the control group who received text messages unrelated to quitting. At 6-months abstinence was significantly increased in the intervention group versus the control group (10.7% vs. 4.9%; p<0.0001).

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed pregnancy,
* English speaking,
* 18-55 years of age,
* Are in the preparation stage of change and willing to set a quit date within 30 days and before 35 weeks gestation,
* Have a cellular phone that is capable of receiving text messages, and be willing to pay for any related fees for testing.
* Willing and able to commit to the visit schedule

Exclusion Criteria:

* Gestational age > 35 weeks at quit date
* If subjects are in the pre-contemplative or contemplative stages of change or have already received 30 minute pharmacy education targeted for the quit date in this pregnancy.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-03; Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine J Mathews, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Forinash AB, Yancey A, Chamness D, Koerner J, Inteso C, Miller C, Gross G, Mathews K. Smoking Cessation Following Text Message Intervention in Pregnant Women. Ann Pharmacother. 2018 Nov;52(11):1109-1116. doi: 10.1177/1060028018780448. Epub 2018 Jun 1. PMID 29857773

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 patient were randomized to the texting group and 26 to the control. However, 9 in the texting group and 10 in the controls did not follow up for any study procedures of data collection, so we do not have data to report on them.
Period: Overall Study
Arm/Group | Texting Group | Control Group
Started | 23 | 26
Completed | 14 | 16
Not Completed | 9 | 10
Not completed — Withdrawal by Subject | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Texting Group | Control Group | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 13 | 23
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Carbon Monoxide Levels
Description: self-reported cessation rates at 1 month, as verified by exhaled carbon monoxide levels
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Texting Group | Control Group
Number analyzed (Participants) | 14 | 16
Participants | 8 | 5

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Texting Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

LIMITATIONS AND CAVEATS:
Due to challenges with recruitment and retention, the study was underpowered to detect statistical differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT03024606/Prot_SAP_000.pdf